CLINICAL TRIAL: NCT04988425
Title: Subcutaneous Injection of TNFα Monoclonal Antibody for Treating Traumatic Acute Spinal Cord Injury
Brief Title: TNFα Monoclonal Antibody for Acute Spinal Cord Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: The First People's Hospital of Kunshan (Other); Traditional Chinese Medicine Hospital of Kunshan, China (Unknown); 904th Hospital of the Joint Logistics Support Force of the PLA (Other); The Sixth People's Hospital of Nantong, China (Unknown); Zhejiang Provincial Hospital of TCM (Other)
Responsible Party: Principal Investigator, Xuhua Lu, Director of Traumatic Orthopaedic Department, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021070701
Record Dates: First submitted 2021-07-07; First posted 2021-08-03 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Masking Description: Random grouping
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TNFα monoclonal antibody group (Experimental): Subcutaneous injection of 50mg of TNFα monoclonal antibody immediately after admission before surgery.
  Interventions: Drug: TNFα Monoclonal Antibody
- Methylprednisolone group (Active Comparator): Injection of 500mg of methylprednisolone immediately after admission before surgery.
  Interventions: Drug: Methylprednisolone
- Control group (Placebo Comparator): Injection of the same volume of saline immediately after admission before surgery.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: TNFα Monoclonal Antibody — Subcutaneous injection of 50mg of TNFα monoclonal antibody immediately after admission before surgery.
  Arms: TNFα monoclonal antibody group
Drug: Methylprednisolone — Injection of 500mg of methylprednisolone immediately after admission before surgery.
  Arms: Methylprednisolone group
Drug: Saline — Injection of the same volume of saline immediately after admission before surgery
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of subcutaneous injection of TNFα monoclonal antibody cells for the treatment of traumatic acute spinal cord injury. Spinal cord injury can be divided into three phases, which are acute (within 2 weeks), sub-acute (2 weeks to 6 months), and chronic (over 6 months). The pathological process of spinal cord injury include primary injury (initial traumatic insult) and a progressive secondary injury cascade characterized by ischemia, proapoptotic signaling, peripheral inflammatory cell infiltration and the release of proinflammatory cytokines. Secondary injury plays a key role in the loss of spinal cord function after trauma. So early treatment to prevent the secondary injury is the key to improve prognosis. TNFα monoclonal antibody is a TNF-α inhibitor that could control inflammatory response, and now widely used in the treatment of Ankylosing spondylitis, Rheumatoid arthritis and other autoimmune diseases. In this study, the investigators will treat patients with acute spinal cord injury with TNFα monoclonal antibody and compare with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 60 years
* Traumatic spinal cord injury
* ASIA Impairment Scale A-D
* The injury must be within two weeks
* Patients submitted written informed consent

Exclusion Criteria:

* Traumatic spinal cord injury with brain injury or peripheral nerve injury
* Patients with severe multiple injuries and unstable vital signs
* Non-traumatic spinal cord injury caused by spinal tumors, hematoma, myelitis, etc.
* Patients with central spinal cord injury
* Patients with a completely transected spinal cord
* Patients with fever or acute infection
* Ongoing infectious disease, such as tuberculosis, HIV, hepatitis, syphilis, etc.
* Patients with malignant tumour
* Patients with neurodegenerative diseases, or any neuropathies
* Patients with ankylosing spondylitis
* Patients with a previous history of spinal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
American Spinal Injury Association Impairment Scale(ASIA) | baseline, 1 month, 3 months, 6 months and 12 months post-treatment
  Change in sensory and motor function as measured by the American Spinal Injury Association Impairment Scale (ASIA). The scale ranked from A to E, A indicates the the most severe spinal cord injury and E indicates no neurological deficit.

SECONDARY OUTCOMES:
Incidence of adverse events | 1 month post-treatment
  Any abnormal signs, symptoms, findings, or diseases that emerge or worsen relative to baseline in 1 month posttreatment will be recorded as adverse event
Motor Evoked Potentials (MEP) and Somatosensory Evoked Potentials (SSEP) test | baseline, 3 months, 6 months and 12 months post-treatment
  Change in sensory and motor function will be measured by SSEP and MED test
Residual urine test | baseline, 3 months, 6 months and 12 months post-treatment
  Change in residual urine as measured by ultrasound test

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Lu, M.D., Principal Investigator — Shanghai Changzheng Hospotal
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be available through email when requested